CLINICAL TRIAL: NCT05869708
Title: Personalizing Self Neuro-modulation Therapy for Major Depressive Disorder (MDD) With Anhedonia Using Clinical Biomarkers for MDD Subtypes
Brief Title: PRISM Neurofeedback Training for MDD Anhedonic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GrayMatters Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLP011
Record Dates: First submitted 2023-04-23; First posted 2023-05-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anhedonia
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Arm (Experimental): Subjects randomized into the Active arm will receive RS-EFP-NF Prism training as an adjunct to standard of care.
  Interventions: Device: Active RS-EFP
- Control Arm (Sham Comparator): Subjects randomized into the Control arm will receive a Sham-EFP-NF training with the same schedule as the active arm, adjunct to standard of care.
  Interventions: Device: Sham RS-EFP

INTERVENTIONS:
Device: Active RS-EFP — A minimum of 10 and up to 15 active NF Prism training sessions, aimed to train for upregulating the RS activity. Sessions will occur twice a week, on nonconsecutive days, over 5-8 consecutive weeks. Subjects will also receive two single booster sessions, one month and two months after their last training session.
  Arms: Active Arm
Device: Sham RS-EFP — a minimum of 10 and up to 15 sham NF Prism training sessions, aimed to train for upregulating the RS activity. Sessions will occur twice a week, on nonconsecutive days, over 5-8 consecutive weeks. Subjects will also receive two single sham booster sessions, one month and two months after their last training session.
  Arms: Control Arm

SUMMARY:
The goal of this interventional double-blind study is to demonstrate the safety and efficacy of PRISM neurofeedback training within an MDD Anhedonia sample.

The goals of this study include:

1. Demonstrating the safety and efficacy of Prism Neurofeedback training within an MDD Anhedonia sample;
2. Identifying clinical profile/symptoms-based biomarkers (e.g., Hamilton Depression Rating Scale - HDRS-21, Dimensional Anhedonia Rating Scale - DARS, Snaith-Hamilton Pleasure Scale for Clinicians SHAPS) scores that can be used by clinics to administer Prism therapy in conjunction with standard of care (SOC) therapy;
3. Producing initial guidelines for integrating Prism neurofeedback training for MDD therapy with MDD Anhedonia (SOC).

Participants will be randomly assigned to one of two arms, Active, or Sham.

DETAILED DESCRIPTION:
During the study, participants will perform the following:

* Complete clinical assessments using questionnaires, an MRI scan, and tasks that probe reward responsivity, learning, and motivation.
* Perform at least 10 sessions but optimally 15 (+/-3) neurofeedback training sessions (performed twice a week on nonconsecutive days for 5-8 weeks).
* Complete the same clinical assessments, post-NF training MRI scan, and tasks same as in the screening/baseline stage.

Researchers will compare the sham and treatment arm to evaluate if the neurofeedback effect reduced MDD symptoms in MDD patients with Anhedonia.

ELIGIBILITY:
MDD subjects

Inclusion Criteria:

1. Ages 22 to 65
2. Any gender and all ethnic/racial origins
3. Diagnosis of MDD with Anhedonia, established according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5). MDD diagnosis will be determined via the Structured Clinical Interview for DSM-5 (SCID-V) with ≥17 on the Hamilton Depression Rating Scale (HDRS)-211 and ≥25 on the Snaith-Hamilton Pleasure Scale (SHAPS-C)
4. Fluency in written and spoken English
5. Ability to give signed, informed consent either written or electronic (via REDCap eConsent)
6. Normal or corrected-to-normal vision and hearing
7. Ability to adhere to the study schedule

Exclusion Criteria (All Subjects):

Imaging Exclusions 1. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

2. Contraindications to MRI (e.g., metal in the body, claustrophobia). 3. Hairstyles that prevent application of the EEG net (e.g., braids, dreadlocks, cornrows, recently dyed hair) Comorbidity Exclusions

1. A history of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder, organic mental disorder, severe borderline or antisocial personality disorder, current bulimia nervosa2, current binge eating disorder2, or current anorexia nervosa3.
2. Lifetime Diagnosis of autism or intellectual disability at the discretion of the investigator.
3. Current primary diagnosis of posttraumatic stress disorder (PTSD), specific phobia, panic disorder, social anxiety disorder, obsessive compulsive disorder, or generalized anxiety disorder; subjects with MDD as a primary diagnosis may be included.
4. First-degree relatives with a history of psychotic disorder or psychotic symptoms outside of the context of a mood disorder (i.e., MDD or bipolar disorder)
5. Any suicidal behavior in the past 1 year (i.e., actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior) assessed using Columbia -Suicide Severity Rating Scale (C-SSRS) prior to screening and during the screening period.
6. Diagnosis for current moderate or severe substance or alcohol use disorder (SUD/AUD) within the past month (as defined in DSM-5-substance use disorder) with the exception of cocaine or stimulant abuse which will lead to an automatic exclusion.

Additional Substance and Drug Use Exclusions

1. Any current drug use as assessed by a positive result on urine drug test (covering cocaine, opiates, amphetamines, methamphetamines, phencyclidine, MDMA, benzodiazepines, methadone, oxycodone, tricyclic antidepressants, and barbiturates)

   1. Allow positive result for cannabinoids if participant verbally confirms they have not used MJ in past 12 hours prior to study visit
2. Use of any antibiotics in the 24 hours prior to an MRI scan procedure
3. Recent use (within 4 weeks) or any current medication that affects blood flow or blood pressure, or which is vasodilating/vasoconstricting (for participants undergoing neuroimaging) Medical Exclusions

1. Any unstable medical condition, as per the clinical judgement of the investigator.

2. A history of seizures, at risk for seizure (e.g., history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes or familial or personal history of epilepsy) or have been diagnosed with a seizure disorder.

Treatment Exclusions

1. Any prescribed Benzodiazepine which cannot be ceased for the duration of the study (with a washout period of at least 2 weeks prior to the first Prism training session) or which cannot be replaced with short-acting benzodiazepines that are taken only for sleeping during the night at equivalent daily dose of up to 3 mg.
2. History of ECT, TMS, or Ketamine in the current Major Depressive Episode (allowable in previous MDEs)
3. Completion of two full courses of other therapies within the current episode
4. Any psychotropic medication other than a stable dose of antidepressants, e.g., bupropion, selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitor (SNRIs), St. John's Wort, or SAMe.
5. Any change in - or initiation of - fluoxetine within the past 8 weeks or other SSRIs or SNRIs antidepressants, bupropion, simulants, or other psychiatric medications within the past 4 weeks. At the time of recruitment, patients must have no intention of changing their medication or psychotherapy during the study duration.
6. Recent initiation (within the past 2 months) of psychotherapy; continuation of established maintenance supportive therapy will be permitted.
7. Enrollment in another therapeutic clinical study at screening or within 2 months prior to screening or intended enrollment within the duration of this study

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
HDRS-21 | 9 weeks
  The HDRS (also known as the Ham-D) is the most widely used clinician-administered depression assessment scale. It is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. Each item on the questionnaire is scored on a 3- or 5-point scale, depending on the item, and the total score is compared to the corresponding descriptor. Assessment time is about 20 minutes.

SECONDARY OUTCOMES:
Snaith Hamilton Pleasure Scale - self reported (SHAPS-SR) | 9 weeks
  The Snaith Hamilton Pleasure Scale (Snaith et al., 1995) is a 14- item self-administered measure of anhedonic symptoms. The purpose of this assessment is to evaluate the ability to enjoy/experience pleasure in activities in the past week. Each item is rated on a 4-point Likert scale, where the total score ranges between 0 to 42 and a higher total score means a worse outcome.
HDRS-21 | 3 months
  The HDRS (also known as the Ham-D) is the most widely used clinician-administered depression assessment scale. It is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. Each item on the questionnaire is scored on a 3- or 5-point scale, depending on the item, and the total score is compared to the corresponding descriptor. Assessment time is about 20 minutes.
Snaith Hamilton Pleasure Scale - self reported (SHAPS-SR) | 3 months
  The Snaith Hamilton Pleasure Scale (Snaith et al., 1995) is a 14- item self-administered measure of anhedonic symptoms. The purpose of this assessment is to evaluate the ability to enjoy/experience pleasure in activities in the past week. Each item is rated on a 4-point Likert scale, where the total score ranges between 0 to 42 and a higher total score means a worse outcome.
The clinical global impression (CGI-I) | 9 weeks
  The CGI-I Scale - of Clinical Global Impression (Guy et.al, 1976) - is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Rated within the range of 0 to 7, lower scores indicate improved outcomes while higher scores indicate worsen outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No